CLINICAL TRIAL: NCT05850312
Title: Gamified Digital Intervention to Enhance the Efficacy of Exposure Therapy for OCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-FY2023-154
Record Dates: First submitted 2023-03-03; First posted 2023-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Experimental Video Games; Behavioral Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Round 1 (Experimental): Initially the aim is to recruit 5 clinicians to play the existing MoM game in a controlled environment. The goal is to congregate their collective feedback about the existing game as well as additional features that needs to be implemented to comprise Exposure Therapy to treat OCD with cleanliness. In addition, a feasibility analysis will be conducted to the proposed gameplay described in section 3.1.1. With these assessments, implementation process will be initiated.
  Interventions: Device: Gamified Digital Intervention - Feasibility Analysis on MoM
- Round 2 (Experimental): A second round of data collection will be conducted with a sample size of 10 subjects (5 clinicians and 5 non-clinician adults). In this second round it is intended to recruit both clinicians and non-clinicians as participants of the study. In the first phase of this study, the clinicians will play the game MoMG to carefully review the revised version of the game. In the second phase the non-clinicians will play the game in presence of clinicians with a goal to ensure that this game does not harm and the gameplay is enjoyable to the participants. While recruiting the non clinicians, it will be ensured via screening that none of the the participants have OCD or other germaphobia.
  Interventions: Device: Gamified Digital Intervention

INTERVENTIONS:
Device: Gamified Digital Intervention - Feasibility Analysis on MoM — In first round we aim to clinically analyze the game Militant of the Maze (MoM) as a vehicle for Exposure Theory, including, play, observation, and feedback from five clinicians.
  Arms: Round 1
Device: Gamified Digital Intervention — In the first phase of round 2 of the study, 5 clinicians will play the game to evaluate the revised game MoMG. In the next phase, 5 carefully-selected non-clinician participants will play the game. under real-time observation of clinicians, to ensure that subjects experience no harm, and that the gameplay is interesting and enjoyable.
  Other Names: Gamified Digital Intervention - Analyzing MoMG
  Arms: Round 2

SUMMARY:
Aim 1 - Clinically analyze the game Militant of the Maze (MoM) as a vehicle for Exposure Theory, including, play, observation, and feedback from five clinicians. MoM, developed in our lab, emphasizes the significance of controlled alternation, while achieving a goal of an individual suffering from OCD who considers that there is only one optimal way of solving a problem. Since this game is already developed in the PI's research lab, this can accommodate OCD treatment strategies, a significant amount of time can be conserved. While the game runs on hand-held devices, all proposed subject testing will be conducted in the laboratory.

Aim 2: Based on the feedback, modifications will be made in MoM to inject narrative, mechanics, and gameplay to address the features of Exposure Therapy that aims to deal with the ob- session/compulsion of cleanliness. One of the key mechanisms of this game will be exposing the patients to simulated human sneezing by using animated splashes of droplets on the screen that the patent will need to wipe without becoming agitated.

Aim 3: Once the game is developed, another round of laboratory case study will be conducted. In the first phase of this round of study, 5 clinicians will play the game to evaluate the revised game MoMG. In the next phase, 5 carefully-selected non-clinician participants will play the game. under real-time observation of clinicians, to ensure that subjects experience no harm, and that the gameplay is interesting and enjoyable. Observational data, including stress measures such as real- time heart rate will be collected, along with verbal protocol and video recording for further analysis, game enhancement, and testing as an exposure therapy mechanism.

DETAILED DESCRIPTION:
A laboratory experiment will be conducted to analyze the playability and feasibility of the proposed game as an effective tool of Exposure Therapy to treat people with cleanliness OCD. The experimental procedure will include the following 3 steps-

1. Initially the aim is to recruit 5 clinicians to play the existing MoM game in a controlled environment. The goal is to congregate their collective feedback about the existing game as well as additional features that needs to be implemented to comprise Exposure Therapy to treat OCD with cleanliness. In addition, a feasibility analysis will be conducted to the proposed gameplay. With these assessments, implementation process will be initiated.
2. A newer and updated version of the game MoM will be implemented based on the outcome of the analysis conducted in the first phase of this experiment. Upon the completion of the development procedure several test runs will be operated to ensure the playability and quality of the game.
3. A second round of data collection will be conducted with a sample size of 10 subjects. In this second round in is intended to recruit both clinicians and non-clinicians as participants of the study. While recruiting, it will be ensured none of the the participants have OCD or other germaphobia. This experiment as well will be conducted in a controlled environment with a goal to ensure that this game does not harm any individual and the gameplay is enjoyable. Data will be collected through various media. Players' certain actions and interactions (e.g. cognitive pause) will be logged in the back end during the gameplay. After certain gameplay, the players' will be provided survey questionnaires, which will long their positive and negative experience and the intrinsic motivation of the gameplay. In addition, to avoid any bias, observational data will be logged through video recording.

ELIGIBILITY:
Inclusion Criteria:

* Must be a clinician (for Group 1)
* Must be an adult with no symptom of OCD/phobia (for Group 2)

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Measuring the heart rate control of the player | 2-3 months
  A measurement of heart rate of the player will be recorded during the gameplay of MoM
Measuring Game Experience Questionnaire (GEQ) | 2-3 months
  The Game Experience Questionnaire (GEQ) was designed by IJsselsteijn et al. in 2013 to assess the game experience of an individual. This questionnaire comprises three modules: The Core Questionnaire, The Social Presence Module, and The Post-game Module. The evaluation of the game experience is done based on seven components: Immersion, Flow, Competence, Positive and Negative Affect, Tension, and Challenge. It contains 33 questions in total for all seven elements Each question is associated with a 5-point Likert scale where 0 represents not at all and 4 signifies extremely. For this experiment, only Immersion, Flow, Challenge, Positive Affect, and Negative Affect have been considered
Measuring Intrinsic Motivational Inventory (IMI) | 2-3 months
  The Intrinsic Motivation Inventory (IMI) is a constructive measurement system to assess an individual's subjective experience related to a target activity in laboratory experiments. Through this, it is possible to assess 7 sub-scales: Interest/Enjoyment, Perceived Competence, Effort/Importance, Pressure/Tension, Perceived Choice,Value/Usefulness, and Relatedness. Each subscale consists of a number of statements. One can respond to the subscales on a scale of 1 to 7 where 1 is not at all true and 7 signifies very true. For this experiment, only the level of Interest/Enjoyment, Perceived Competence, Effort/Importance, and Pressure/Tension were observed

CONTACTS AND LOCATIONS:
Overall Officials: Farjana Z Eishita, PhD, Principal Investigator — Assistant Professor

IPD SHARING:
Plan to Share IPD: Undecided
Once the study is completed data analysis will be conducted and then the decision will be made based on the outcome.

REFERENCES:
- [Background] Gavin Andrews. Clinical handbook of psychological disorders: a step-by-step treatment manual (4th edn) edited by david h. barlow. guilford press. 2007. 689pp. isbn: 9781593855727. The British Journal of Psychiatry, 194(5):473-473, 2009.
- [Background] David H Barlow. Clinical handbook of psychological disorders: A step-by-step treatment manual. Guilford publications, 2021.
- [Background] T Atilla Ceranoglu. Video games in psychotherapy. Review of General Psychology, 14(2):141-146, 2010.
- [Background] Rachel K Chesham, John M Malouff, and Nicola S Schutte. Meta-analysis of the efficacy of virtual reality exposure therapy for social anxiety. Behaviour Change, 35(3):152-166, 2018.
- [Background] Fleming TM, Bavin L, Stasiak K, Hermansson-Webb E, Merry SN, Cheek C, Lucassen M, Lau HM, Pollmuller B, Hetrick S. Serious Games and Gamification for Mental Health: Current Status and Promising Directions. Front Psychiatry. 2017 Jan 10;7:215. doi: 10.3389/fpsyt.2016.00215. eCollection 2016. PMID 28119636
- [Background] Julian Frommel, Martin Dechant, and Regan Mandryk. The potential of game streaming as exposure therapy for social anxiety. Proc. ACM Hum.-Comput. Interact., Vol. 5, No. CHI PLAY,, 2021.
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Granic I, Lobel A, Engels RC. The benefits of playing video games. Am Psychol. 2014 Jan;69(1):66-78. doi: 10.1037/a0034857. Epub 2013 Dec 2. PMID 24295515
- [Background] Ho CS, Chee CY, Ho RC. Mental Health Strategies to Combat the Psychological Impact of Coronavirus Disease 2019 (COVID-19) Beyond Paranoia and Panic. Ann Acad Med Singap. 2020 Mar 16;49(3):155-160. No abstract available. PMID 32200399
- [Background] Horne-Moyer HL, Moyer BH, Messer DC, Messer ES. The use of electronic games in therapy: a review with clinical implications. Curr Psychiatry Rep. 2014 Dec;16(12):520. doi: 10.1007/s11920-014-0520-6. PMID 25312026
- [Background] Krzyszkowiak W, Kuleta-Krzyszkowiak M, Krzanowska E. Treatment of obsessive-compulsive disorders (OCD) and obsessive-compulsive-related disorders (OCRD). Psychiatr Pol. 2019 Aug 31;53(4):825-843. doi: 10.12740/PP/105130. Epub 2019 Aug 31. English, Polish. PMID 31760412
- [Background] Lau HM, Smit JH, Fleming TM, Riper H. Serious Games for Mental Health: Are They Accessible, Feasible, and Effective? A Systematic Review and Meta-analysis. Front Psychiatry. 2017 Jan 18;7:209. doi: 10.3389/fpsyt.2016.00209. eCollection 2016. PMID 28149281
- [Background] Liu W, Zhang H, He Y. Variation in Obsessive-Compulsive Disorder Symptoms and Treatments: A Side Effect of COVID-19. Int J Environ Res Public Health. 2021 Jul 12;18(14):7420. doi: 10.3390/ijerph18147420. PMID 34299871
- [Background] Regan L Mandryk, Max V Birk, Adam Lobel, Marieke van Rooij, Isabela Granic, and Vero Van- den Abeele. Games for the assessment and treatment of mental health. In Extended Abstracts Pub- lication of the Annual Symposium on Computer-Human Interaction in Play, pages 673-678. ACM, 2017.
- [Background] McKay D, Minaya C, Storch EA. Conducting exposure and response prevention treatment for contamination fears during COVID-19: The behavioral immune system impact on clinician approaches to treatment. J Anxiety Disord. 2020 Aug;74:102270. doi: 10.1016/j.janxdis.2020.102270. Epub 2020 Jul 1. PMID 32650220
- [Background] Ornell F, Braga DT, Bavaresco DV, Francke ID, Scherer JN, von Diemen L, Kessler FHP. Obsessive-compulsive disorder reinforcement during the COVID-19 pandemic. Trends Psychiatry Psychother. 2021 Apr-Jun;43(2):81-84. doi: 10.47626/2237-6089-2020-0054. Epub 2021 Jan 22. PMID 33503168
- [Background] Pandita S, Mishra HG, Chib S. Psychological impact of covid-19 crises on students through the lens of Stimulus-Organism-Response (SOR) model. Child Youth Serv Rev. 2021 Jan;120:105783. doi: 10.1016/j.childyouth.2020.105783. Epub 2020 Dec 5. PMID 33518862
- [Background] Rus-Calafell M, Gutierrez-Maldonado J, Botella C, Banos RM. Virtual reality exposure and imaginal exposure in the treatment of fear of flying: a pilot study. Behav Modif. 2013 Jul;37(4):568-90. doi: 10.1177/0145445513482969. Epub 2013 Apr 12. PMID 23585557
- [Background] Suso-Ribera C, Fernandez-Alvarez J, Garcia-Palacios A, Hoffman HG, Breton-Lopez J, Banos RM, Quero S, Botella C. Virtual Reality, Augmented Reality, and In Vivo Exposure Therapy: A Preliminary Comparison of Treatment Efficacy in Small Animal Phobia. Cyberpsychol Behav Soc Netw. 2019 Jan;22(1):31-38. doi: 10.1089/cyber.2017.0672. Epub 2018 Oct 18. PMID 30335525
- [Background] Rifat Ara Tasnim and Farjana Z Eishita. Mom an effort to comprising cbt in digital gaming. In 2020 IEEE 8th International Conference on Serious Games and Applications for Health (SeGAH), pages 1-8. IEEE, 2020.
- [Background] NAUvais.Obsessive-compulsivedisorderfollowingcovid-19infection.ThePrimaryCareCompanion for CNS Disorders, 23(6):38521, 2021.